CLINICAL TRIAL: NCT03107351
Title: Validation Study of Cardiac Linear and Torsional Contractility Measurements With a New Technology: Multi Dimensional Kineticardiography (MKCG)
Brief Title: Cardiac Linear and Torsional Contractility Measurements With a New Technology: Multi Dimensional Kineticardiography
Acronym: MultiKinVal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Philippe Van de Borne, Professor, Erasme University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: P2016/474
Record Dates: First submitted 2017-02-22; First posted 2017-04-11 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Double blind randomized crossover active vs placebo
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repeatability measures (Sham Comparator): In this arm, healthy subjects will undergo repeated measures at different times of the day.
  Interventions: Device: Cardiac assessment repeatability with Kino-cardiograph
- Contractility changes measures (Experimental): In this arm, healthy subjects will have their cardiac contractility increased in a controlled way and assessed with both HK and echocardiography.
  Interventions: Device: Cardiac contractility assessments with Kino-cardiograph

INTERVENTIONS:
Device: Cardiac contractility assessments with Kino-cardiograph — Cardiac contractility will be assessed with Kino-cardiograph device. Echocardiography will also be used for the experimental arm
  Arms: Contractility changes measures
Device: Cardiac assessment repeatability with Kino-cardiograph — Cardiac contractility will be assessed with Kino-cardiograph device only, at different times of the day to assess the repeatability of the measures.
  Arms: repeatability measures

SUMMARY:
This study aims to validate the possibility to track cardiac contractility changes with a new technology called 'Heart Kinetic' (HK). HK measurements will be realized and compared echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 50 years old.
* Healthy without medical cardiac conditions history.
* Non smoker.
* Does not take any drugs or medications.
* Does not participate in other clinical study or trial.
* BMI (Body Mass Index) in between 20 and 25 kg/m2.

Exclusion Criteria:

* Being younger than 18 or older than 50 years old.
* Having had previous cardiac conditions or present disease.
* Being a regular smoker.
* Taking any drugs or medications
* Taking part in another clinical study or trial.
* BMI (Body Mass Index) lower than 20 or higher than 25 kg/m2.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
HK reproducibility validation | day 1
  Validate the reproducibility of HK measurements in a clinical environment.
Cardiac contractility tracking with HK | day 1
  Proof that the HK technology can track physiological cardiac changes while comparing with gold standard echocardiography and inducing a cardiac contractility change with dobutamine infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Erasme, Brussels, Anderlecht, Belgium

REFERENCES:
- [Derived] Hossein A, Rabineau J, Gorlier D, Pinki F, van de Borne P, Nonclercq A, Migeotte PF. Effects of acquisition device, sampling rate, and record length on kinocardiography during position-induced haemodynamic changes. Biomed Eng Online. 2021 Jan 6;20(1):3. doi: 10.1186/s12938-020-00837-5. PMID 33407507